CLINICAL TRIAL: NCT02757937
Title: Study to Measure Merck Engage Usability and Conduct Outcomes Testing
Brief Title: Reaching Better Health Study: A Website to Improve Type 2 Diabetes Self-Management
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-011892
Record Dates: First submitted 2016-04-25; First posted 2016-05-02 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Medication Adherence; Self-efficacy; Behavior; Diabetes; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence; Behavior; Diabetes Mellitus | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health & Wellness Website (Experimental): Subjects will receive access to an interactive health & wellness website for 6 months. The site aims to provide patients with information, tools, and resources to manage their chronic condition (e.g., Type 2 diabetes). The website will send subjects emails with tips to help them take better care of their diabetes, such as how to track diet and exercise habits and how to cook healthy meals. The study researchers will keep track of how many times subjects access the website and which parts of the site are most commonly viewed. Intervention subjects will receive questionnaires assessing engagement and satisfaction with the website. Subjects will also complete questionnaires at baseline and 2, 4, and 6 months post-baseline.
  Interventions: Behavioral: Health & Wellness Website
- Control Arm (Other): Subjects in the control arm will continue with standard diabetes care without getting access to the intervention website. Subjects will also complete questionnaires at baseline and 2, 4, and 6 months post-baseline. Control subjects will be granted access to the health & wellness website after the study is completed.
  Interventions: Other: Control Arm

INTERVENTIONS:
Behavioral: Health & Wellness Website — Educational website for patients with chronic disease (i.e., Type 2 diabetes, asthma, high blood pressure, high cholesterol). The website is a free interactive resource to help patients manage their health condition(s) each day and to help them achieve their goals. It is a multichannel health and wellness platform to help patients adhere to their treatment and care plans between office visits.
  Arms: Health & Wellness Website
Other: Control Arm — Continue with standard diabetes care without getting access to the intervention website.
  Arms: Control Arm

SUMMARY:
Diabetes is one of the most common chronic illnesses among adults in the United States. Internet-based interventions and health promotion websites for patients with Type 2 Diabetes are typically low-cost, easily accessible, and attractive. The purpose of this study is to determine whether participants' utilization of a health & wellness website focused on diabetes self-management increases participants' self-reported self-efficacy toward managing their Type 2 Diabetes through behavior change and self-reported medication adherence compared to standard care.

DETAILED DESCRIPTION:
Diabetes is one of the most common chronic illnesses among adults in the United States. Merck & Co., Inc. has produced an innovative website to engage adult patients in chronic illness self-management and medication adherence. Internet-based interventions and health promotion websites for patients are typically low-cost, easily accessible, and attractive. However, there is a growing need for improved measurement, implementation and evaluation of online health interventions to ensure patient engagement and produce more significant behavior change that can impact patients' health over the long term.

The primary objective of this study is to determine whether utilization of the health and wellness website increases participants' self-reported self-efficacy toward managing their Type 2 Diabetes through behavior change and self-reported medication adherence.

This study comprises a randomized controlled trial utilizing the website as the self-management support intervention. There is no interventional medical treatment, and no change in patients' medical care. In collaboration with University of Pennsylvania, potential participants will be identified and recruited from the Penn Medicine outpatient population based on specific inclusion/exclusion criteria. Participants will remain in the study for 6 months.

Participants will be randomly assigned to the intervention or control condition (no exposure). Those in the intervention arm will have access to health & wellness website for nine months post enrollment. Online surveys will be delivered during this nine month period. Primary outcomes will be baseline-to-two month and baseline-to-4 month changes in diabetes management self-efficacy scores as measured by the Diabetes Self-Efficacy Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a current patient in the Penn Medicine outpatient healthcare system
* Patient's Primary Care Physician (PCP) or Endocrinologist is a Penn Medicine provider
* Patient has a 12 month history of healthcare utilization in the Penn Medicine system (in-office PCP/endocrinologist visits)
* Patient has complete data (ICD-10 code for Type 2 diabetes diagnosis, date of diagnosis, name and mailing address information) in the Penn Data Warehouse
* Patient is diagnosed with Type II Diabetes as indicated by ICD-10 Codes: E11.** (including any newly diagnosed)
* Patients' HbA1c was ≥8.0% in last 6 months (if more than one A1c result present in record, most recent measurement assessed)
* Patient can read and understand English well enough to complete study tasks.
* Patient has regular access to a telephone
* Patient has at least bi-weekly access to internet and email
* Patient agrees to release their medical record information to Children's Hospital of Philadelphia research team

Exclusion Criteria:

* Patient is deceased
* Patient has indicated "Do Not Solicit for Research" in medical record
* Patient is less than 18 years of age
* Patient is older than 75 years old
* Patient uses an insulin pump or injectable insulin to treat/manage their diabetes.
* Patient is non-English speaking
* Patient does not have HbA1c% in chart from last 6 months
* Patients' HbA1c in last 6 months is <8.0%
* Patient is currently taking medications that can raise glucose levels, such as steroids
* Patient has a history of cognitive disorders, mental illness, and/or cognitive impairment that may impact their ability to use an online website, including, dementia, Alzheimer's disease, Parkinson's disease, traumatic brain or head injury, and psychosis
* Patient has history of Heart Failure (included Chronic Heart Disease, Chronic Heart Failure) and/or Chronic Kidney Disease, and has had other serious cardiovascular conditions (e.g, heart attack or stroke) in the last 6 months
* Patient has history of endocrine gland cancers or pancreatic cancers
* Patient is undergoing chemotherapy or immunotherapy treatment in last 6 months
* Patient's medical record contains ICD-10 Code for Type I diabetes diagnosis.
* Patient's medical record contains ICD-10 Code for pregnancy-related diabetes:

  * 024.419 (gestational diabetes)
  * 024.419 (antepartum gestational diabetes)
  * Z79.4 (type II long term insulin use)
  * 024.91x (pregnant women who are diabetic)
* Patient is Pre-diabetic or borderline Type 2 diabetic
* Patient is pregnant or lactating
* Patient's electronic medical history data is not available through Penn Medicine's electronic medical record and/or is not complete in Penn Data Store
* Patients who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes Self-Efficacy Scale Score from Baseline to 4 Months | Baseline to 4 months
  The validated Diabetes Self-Efficacy Scale (Lorig et al., 2009) assesses how confident one is in doing certain activities related to diabetes management. There are 8 items in this measure with each one pertaining to a different activity. Each item is rated on a continuous scale of 1 to 10, 1 being not at all confident and 10 being totally confident. The score for each item is the number circled and higher value score indicates greater self-efficacy.

SECONDARY OUTCOMES:
Change in Diabetes Knowledge Test Score from Baseline to 4 Months | Baseline to 4 months
  This is a 14 item assessment, measuring general diabetes knowledge, was validated among Type 1 and Type 2 adult diabetics, Cronbach's α = 0.71. Each item is a multiple choice question, with options A-D. For scoring, the total number of questions answered correctly is calculated. The higher the score on the test, the greater knowledge one has about diabetes.
Change in Self-Efficacy Scale Score for Managing Chronic Disease from Baseline to 4 Months | Baseline to 4 Months
  This measure assesses how confident one is when performing various activities related to chronic disease management. There are 6 items on this scale with each one pertaining to a different activity. Each item is rated on a continuous scale of 1 to 10, with 1 being not at all confident and 10 being totally confident. The overall score for the measure is the average value of all the items. A higher score indicates a greater self-efficacy.
Change in glycated haemoglobin (HbA1c) from Baseline to 6 Months | Baseline to 6 Months
  By measuring glycated haemoglobin (HbA1c), clinicians are able to get an overall picture of what average blood sugar levels have been over a period of weeks/months. For people with diabetes this is important as the higher the HbA1c, the greater the risk of developing diabetes-related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Fleisher, PhD, MPH, Principal Investigator — Children's Hospital of Philadelphia

IPD SHARING:
Plan to Share IPD: No